CLINICAL TRIAL: NCT06740084
Title: African Youth in Mind (Y-MIND) - Pilot Feasibility Trial of a Brief Psychological Intervention for Older Adolescents with Depression Delivered Through Senior High Schools in Navrongo, Ghana
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Zimbabwe (Other); University of Ghana (Other); Kamuzu University of Health Sciences (Other); Navrongo Health Research Centre, Ghana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR/DP-23/24-38948; NIHR133384 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Depression Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): Enhanced Usual Care (EUC): Guidance and counselling coordinators in the schools provide some counselling to students who need it. Building on the existing structure, enhanced usual care in the Y-MIND programme, will be enhanced in three ways 1) Teaching staff will receive basic training on common mental health conditions affecting youth in Ghana with an emphasis on depression and suicidal symptoms and treatment. 2) Nurses in all schools and other relevant local health care professionals will be trained in mental health, substance-use and self-harm including guidelines on when and where to refer young people for psychiatric care. 3) The study team will provide a letter for the Guidance and Counselling Coordinators for the participant.
  Interventions: Other: Enhanced Usual Care
- Y-MIND Intervention (Experimental): All participants in the intervention arm will receive the EUC plus the Y-Mind intervention. Y-Mind intervention will be delivered by trained and supervised Guidance and Counselling Coordinators (GCC) at schools in 6 sessions. The six sessions will include a) psychoeducation on depression, b) behavioural activation (helping the participant see the connection between their behaviour, daily activities, and low mood and activity scheduling) and c) problem-solving therapy (the GCC helps the participant identify and define a specific problem to work on, evaluate the potential solutions to the problem, and carry out the selected solution(s)).
  Interventions: Behavioral: Y-MIND Intervention

INTERVENTIONS:
Behavioral: Y-MIND Intervention — All participants in the intervention arm will receive the EUC plus the Y-Mind intervention. Y-Mind intervention will be delivered by trained and supervised Guidance and Counselling Coordinators (GCC) at schools in 6 sessions. The six sessions will include a) psychoeducation on depression, b) behavioural activation (helping the participant see the connection between their behaviour, daily activities, and low mood and activity scheduling) and c) problem-solving therapy (the GCC helps the participant identify and define a specific problem to work on, evaluate the potential solutions to the problem, and carry out the selected solution(s)).
  Arms: Y-MIND Intervention
Other: Enhanced Usual Care — Enhanced Usual Care (EUC): Guidance and counselling coordinators in the schools provide some counselling to students who need it. Building on the existing structure, enhanced usual care in the Y-mind programme, will be enhanced in three ways: 1) Teaching staff will receive basic training on common mental health conditions affecting youth in Ghana with an emphasis on depression and suicidal symptoms and treatment. The WHO guidelines for school health services will form the basis for the training for teachers. 2) Nurses in all schools and other relevant local health care professionals will be trained in mental health, substance-use and self-harm including guidelines on when and where to refer young people for psychiatric care. The World Health Organization (WHO) Mental Health Gap intervention guide (mhGAP) will be used for training of nurses and other health care professionals . 3) The study team will provide a letter for the Guidance and Counselling Coordinators for the participant.
  Arms: Enhanced Usual Care

SUMMARY:
The overarching aim of this pilot study is to assess the feasibility of implementing a psychological intervention (Y-MIND), delivered by school guidance and counselling coordinators, for the treatment of depression among adolescents in senior high schools in Ghana. The study is a parallel arm cluster randomised controlled pilot trial. We will recruit adolescents aged 15 to 18 years in senior high schools. Participants will be randomised to receive the Y-MIND psychological intervention or enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 15 to 18 years in senior high schools located within the Kassena-Nankana Municipality and Kassena-Nankana West District
* Have scored 10 or more on the locally validated Patient Health Questionnaire-9 (PHQ-9)
* be willing and able to be followed up for 5 months and provide informed consent or assent
* For adolescents 15-17 years participants must have 5) access to a caregiver to obtain informed consent
* All participants must have the ability to read, write and communicate in English language.

Exclusion Criteria:

* are currently receiving any psychological treatment (talking therapy) for any common mental disorder through formal health care services
* have active bipolar disorder or psychosis (assessed through a brief screening tool for bipolar disorder and psychosis)
* have advanced or chronic physical illness (assessed through self-report)
* have significant visual or hearing impairment which would interfere with their ability to take part in the study
* are actively suicidal (assessed through the use of a four-item screening tool administered by a psychiatric nurse and reviewed by the trial clinical psychologist

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | At the end of treatment (week 6) (or at their 5 months post baseline assessment if the treatment sessions were not attended)
  Feasibility of the intervention will be measured using the 'Feasibility of Intervention Measure' (FIM) with adolescents who received the Y-MIND intervention.
Symptoms of depression | 5 months post baseline assessment
  Symptoms of depression at 5 months post baseline assessment measured as the difference in mean score on the Patient Health Questionnaire-9 (PHQ-9) between the two arms. Difference in mean PHQ-9 would likely constitute a primary outcome in a later larger definitive trial.

SECONDARY OUTCOMES:
Acceptability and appropriateness of the intervention | At end of Y-MIND intervention sessions or at 5 months post baseline assessment
  Acceptability and appropriateness of the intervention will be measured using the Intervention Appropriateness Measure (IAM), Acceptability of Intervention Measure (AIM) with adolescents at the end of their last intervention session (or at their 5 month post baseline assessment if the intervention session was not attended), and with Guidance and Counselling Coordinators at schools after they have finished delivering all intervention sessions.
  Acceptability will also be explored through interviews with adolescents (at end of 5 months post baseline assessment) and focus group discussions with Guidance and Counselling Coordinators (after they have finished delivering all intervention sessions) to elicit feasibility, acceptability, appropriateness and barriers and or enablers that may influence the effectiveness of the intervention.
Feasibility of the intervention (Guidance and Counselling Coordinators) | At the end of treatment delivery
  Feasibility of the intervention from the perspective of the Guidance and Counselling Coordinators, will also be measured using the Feasibility of Intervention Measure (FIM) with Guidance and Counselling Coordinators.
Fidelity to delivering the psychological intervention | From the first treatment session (week 1) to the end of treatment (week 6)
  Fidelity to delivering the psychological intervention, defined as the extent to which the intervention was delivered as intended, and measured by rating 20% of randomly selected audio-recorded psychological intervention sessions in the experimental arm using a culturally adapted form of ENACT called the 'Problem-Solving Therapy Fidelity Scale (PROOF)' tool.
Symptoms of anxiety | 5 months post baseline assessment
  Symptoms of anxiety at 5 months post baseline assessment measured as the difference in mean score on the General Anxiety Disorder scale (GAD-7) between the two arms.
Alcohol use | 5 months post baseline assessment
  Alcohol use measured as the difference in mean score on the Alcohol Use Disorders Identification Test (AUDIT)

OTHER OUTCOMES:
Feasibility of conducting a fully powered trial | Screening to 5 months post baseline assessment
  Feasibility of conducting a fully powered trial measured as the proportion of those screened who are eligible, the proportion of those eligible who consent to take part, and the proportion of those who consent who complete the 5 month primary follow up assessment.
Resource use and cost of the Y-MIND psychological intervention | Baseline to 5 month post baseline assessment
  Two types of resource use and cost data will be collected for the economic evaluation; patient and programme level costing of both direct (healthcare cost) and indirect (productivity loss) cost. Both financial (actual money spent) and economic cost (e.g. donated items and volunteering time) will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Navrongo Health Research Centre, Navrongo, Ghana

REFERENCES:
- [Derived] Jopling R, Attah D, Abas M, Adde KS, Goldsmith K, Bere T, Nyamayaro P, Aborigo RA, Barrett B, Owusu L, Glozah F, Akanlu A, Bawa S, Achana FS, Danese A, Smith P, Seward N, Kumwenda M, Chibanda D, Weobong B. African Youth in Mind - Protocol of a Pilot feasibility trial of a brief psychological Intervention for older adolescents with depression delivered through senior high schools in Navrongo, Ghana. PLoS One. 2025 Apr 1;20(4):e0319462. doi: 10.1371/journal.pone.0319462. eCollection 2025. PMID 40168302